CLINICAL TRIAL: NCT05749302
Title: Application of Al18F-NOTA-FAPI PET/CT in Malignant Tumors Expressing Fibroblast-activated Proteins
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NCC3682
Record Dates: First submitted 2023-02-19; First posted 2023-03-01 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Malignancy
Keywords: malignant tumors expressing fibroblast-activated proteins
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Al18F-NOTA-FAPI PET/CT (Experimental): Al18F-NOTA-FAPI PET/CT will be performed on patients with suspected or clearly diagnosed FAP positive-expressing tumors. The patients were injected with Al18F-NOTA-FAPI and underwent PET/CT scan 20~40min after the injection.
  Interventions: Drug: Al18F-NOTA-FAPI

INTERVENTIONS:
Drug: Al18F-NOTA-FAPI — Al18F-NOTA-FAPI was injected into the patients before the PET/CT scans
  Other Names: 18F-FAPI

SUMMARY:
This is an open-label whole-body PET/CT study for investigating the value of Al18F-NOTA-FAPI PET/CT in patients with malignant tumors expressing fibroblast-activated proteins

DETAILED DESCRIPTION:
Tumour tissue includes tumour cells as well as stromal cells (vascular cells, inflammatory cells, fibroblasts etc.). Activated fibroblasts are present not only in tumours but also in wound healing and diseases with stromal remodelling, such as chronic inflammation, myocardial infarction and liver and lung fibrosis.There is a correlation between FAP expression and tumour microvascular density and FAP expression is strongly associated with poor prognosis in a variety of tumours (e.g. colon, pancreatic, ovarian and hepatocellular carcinoma).Over 90% of FAP-positive cancer-associated fibroblasts are found in epithelial tumours, whereas fibroblasts in normal tissues rarely or even do not express FAP, making FAP a potential target for imaging and treatment of various malignancies.

Al18F-NOTA-FAPI is a posionuclide 18F-labelled tumour developer targeting FAP. Current domestic and international studies have shown that it has good stability and high FAP specificity, and shows excellent imaging quality and tumour detection in tumour-bearing mice and cancer patients, and can be used as a broad-spectrum tumour developer for clinical PET/CT imaging for diagnosis and efficacy assessment of tumour patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected or clearly diagnosed Malignant Tumors Expressing Fibroblast-activated Proteins
* signed written consent.
* Willing and able to cooperate with all projects in this study.

Exclusion Criteria:

* pregnancy;
* breastfeeding;
* any medical condition that in the opinion of the investigator may significantly interfere with study compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-01-08 (Actual); Primary Completion 2025-03-08 (Estimated); Study Completion 2026-01-08 (Estimated)

PRIMARY OUTCOMES:
Diagnostic value | through study completion, an average of 1 year
  Sensitivity and Specificity of Al18F-NOTA-FAPI PET/CT for Malignant Tumors Expressing Fibroblast-activated Proteins

CONTACTS AND LOCATIONS:
Overall Officials: Rong Zheng, M.D., Study Director — National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences and PUMC
Locations (1):
- National Cancer Center/Cancer Hospital,Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Chao Yang, China

IPD SHARING:
Plan to Share IPD: No